CLINICAL TRIAL: NCT01065584
Title: An Observational Study to Assess the Effect of Calcineurin Inhibitors on Markers of Transplant Tolerance
Acronym: OSCITT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Armin Goralczyk, Dr., University Medical Center Goettingen
Other Study IDs: OSCITT10
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; Patients undergoing liver transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood cells for fluorescence activated cell sorting and leukocytes for ImmuKnow/Cylex assay
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard immunosuppression: Patients receiving standard immunosuppression after liver transplantation including calcineurininhibitors
- Immunosuppression without calcineurininhibitors: Patients receiving immunosuppression after liver transplantation not based on calcineurininhibitors

SUMMARY:
In experimental and clinical settings it has been shown that transplant tolerance is possible. It has been suggested that regulatory T cells play a beneficial role in the establishment of tolerance. Calcineurin inhibitors may inhibit development of regulatory T cells. However, the influence of calcineurin inhibitors on markers of transplant tolerance has not been studied in patients undergoing liver transplantation. Currently the investigators conduct a study to evaluate the safety and efficacy of a calcineurin inhibitor free immunosuppression in patients undergoing liver transplantation. In this study measurements of immune function and CD4+CD25high-Foxp3+-Il2/CD8+ status will also be performed. In parallel these measurements should be compared to a group of patients undergoing standard immunosuppression including calcineurin inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary liver transplantation
* Patients of age 18 years and older
* Female patients of childbearing potential willing to perform a highly effective contraception during the study and 12 weeks after conclusion of study participation

Exclusion Criteria:

* Multiple organ graft recipients
* Patients receiving ABO incompatible grafts
* Patients with positive cross match
* Pregnancy
* Patients with a psychological, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule
* Patients under guardianship (e.g. individuals who are not able to freely give their informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aiman Obed, Prof. Dr., Study Chair — University Medical Center Goettingen; Armin Goralczyk, Dr., Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Göttingen, Lower Saxony, Germany